CLINICAL TRIAL: NCT01788449
Title: Association of Antibiotic Measures and Control of Bacterial Resistance
Brief Title: Study Evaluating the Association of Antibiotic Measures and Control of Bacterial Resistance
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0910X-101852
Record Dates: First submitted 2009-08-06; First posted 2013-02-11 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Bacterial Infections
Keywords: Antibiotic Bacterial Resistance
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assess efficacy of piperacillin/tazobactam in reducing the cases of colonization and infection of bacteria.

DETAILED DESCRIPTION:
Primarily, this study is designed to assess the efficacy of piperacillin/tazobactam in reducing the cases of colonization and infection of extended-spectrum betalactamases (ESBLs) producing E.coli or K pneumoniae, S aureus methicillin resistant (MRSA) and Enterococcus vancomycin resistant (VRE). Secondly, this study plans to determine the acquisition rate of ESBL producing E Coli or K pneumoniae, methicillin resistant S Aureus (MRSA) and vancomycin resistant Enterococcus spp (VRE), both pre- and post-intervention.

ELIGIBILITY:
All patients admitted in ICU will be enrolled (who qualify for treatment).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intensive Care Unit (ICU)
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2005-05; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Endpoints will be efficacy of piperacillin/tazobactam in reducing colonization rates and infection of E coli or K pneumoniae, vancomycin resistant enterococcus and methicillin resistant S aureus | 8 months

SECONDARY OUTCOMES:
Endpoints will be acquisition and infection rate of ESBL producing E coli or K pneumoniae, vancomycin resistant enterococcus and methicillin resistant S aureus | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer